CLINICAL TRIAL: NCT01104324
Title: Steroid Induced Osteoporosis in the Pediatric Population Ancillary Study- Osteonecrosis in Children With Acute Lymphoblastic Leukemia
Brief Title: Osteonecrosis in Children With Acute Lymphoblastic Leukemia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Halton, Jacqueline, M.D. (Other)
Collaborators: C17 Council (Other)
Responsible Party: Jacqueline Halton MD, Childrens Hospital of Eastern Ontario
Other Study IDs: 08/20E
Record Dates: First submitted 2010-04-12; First posted 2010-04-15 (Estimated); Last update posted 2010-04-15 (Estimated); Status verified 2010-04

CONDITIONS: Osteonecrosis; Acute Lymphoblastic Leukemia
Keywords: bone health; Osteonecrosis; acute lymphoblastic leukemia
MeSH Terms: conditions — Osteonecrosis; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Platlet free plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
Acute lymphoblastic leukemia is the most common form of childhood cancer with current treatment survival rates approaching 80%. Improved outcomes show an increased number of survivors at risk for long-term treatment related side effects including osteonecrosis. Osteonecrosis, or bone death, is caused by blood supply loss to the bone causing pain and poor quality of life. The hips, shoulders, knees and ankles may be affected. Pain is the usual presenting symptom and may become severe requiring surgical decompression or replacement of the affected joint. Long-term effects including arthritis and progressive joint difficulties will not be known for decades. This study aims to determine the risk factors for developing osteonecrosis that will lead to information for earlier detection and prevention. The study will be the basis for future intervention and prevention trials.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in the STOPP-CIS study
* Informed consent of patient or care givers
* >5 years of age at MRI assessment

Exclusion Criteria:

* Individuals with a history of claustrophobia precluding MRI assessment

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with Acute lymphoblastic leukemia who have participated in the STOPP - CIS study will be eligible for this ancillary study.
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2009-07; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
osteonecrosis 1 year post leukemia therapy | One year after completion of therapy for leukemia
  Each participant will undergo MRI of hip, knee, ankle and shoulder to look for ON

SECONDARY OUTCOMES:
Bone mass density and Osteonecrosis | One year post therapy for leukemia
  Is reductions in bone mass density at diagnosis of leukemia associated with the development of ON. These patients are a subset of a lagre study where Bone mass is being measured by DEXA. We will be able to access this data to look for bone mass density
Is Bone loss/failure to accure bone mineral and ON | One year post leukemia therapy
  Is bone loss/failure to accrue bone mineral at a normal rate during chemotherapy is/are associated with the development of ON.These patients are a subset of a lagre study where Bone mass is being measured by DEXA. We will be able to access this data to look for bone loss
Glucocorticoid dose and ON | One year post Leukemia therapy
  Is there a glucocorticoid threshold dose, above which patients are more likely to develop ON. These patients are a subset of a lagre study where glucocorticoid dose is recorded. We will be able to access this data.
Methotrexate dose and ON | One year post leukemia therpy
  Is there a methotrexate threshold dose, above which patients are more likely to develop ON. These patients are a subset of a lagre study where Methotrexate dose is recorded. We will be able to access this data.
Obesity and ON | One year post leukemia therapy
  Is obesity either at diagnosis or during therapy associated with ON. These patients are a subset of a larger group in a larger study. They are recording height weight and BMI. We will be able to access this data.
Weight bearing and non weight bearing activities and ON | One year post leukrmia therapy
  Does weight bearing and non-weight bearing activities play a role in the development of ON. These patients are a subset of a larger study. They are recording these activities. We will be able to use this data.
Hyperlipidemia and On | One year post leukemia therapy
  Is hyperlipidemia associated with the development of ON. Statins (cholesterol lowering medications) have been suggested as a therapeutic intervention to prevent ON. Fasting blood will be tested for lipids at at least one year post chemtherapy.
Thrombophilia and ON | One year post leukemia therapy
  Is thrombophilia associated with the development of ON. Blood will be tested at study entry following one year completion of chemotherapy.Blood will be drawn for protein C, protein S, antithrombin, activated protein C resistance, Factor V Leiden, prothrombin gene complex, MTHFR, lupus anticoagulant and antiphospholipid antibodies and Lipoprotein A.

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Halton, Principal Investigator — Childrens Hospital of Easten Ontario
Locations (10):
- Canada (10):
  - Alberta Children's Hospital, Calgary, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta
  - BC Children's Hospital, Vancouver, British Columbia
  - Winnipeg Children's Hospital, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - Children's Hospital of Western Ontario, London, Ontario
  - Childrens Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Hopital Sainte-Justine, Montreal, Quebec
  - Montreal Children's Hospital, Montreal, Quebec